CLINICAL TRIAL: NCT02616458
Title: The Impact of Ear Pain Anticipatory Guidance Counseling on Otitis Related Visits in a Low Income Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 09-0270
Record Dates: First submitted 2015-11-11; First posted 2015-11-30 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Otitis Media
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ear pain counseling (Experimental): The Ear Pain counseling materials reviewed concepts such as how to recognize ear pain and safely provide pain relief, and how to recognize danger signs that require urgent medical attention. Families were also encouraged to schedule an appointment in the CHC for a possible ear infection rather than going to the emergency department or urgent care facility after hours. The research assistant provided and reviewed proper dosing instructions for acetaminophen and ibuprofen, and provided a prescription for antipyrine/benzocaine analgesic ear drops to each family to use as pain relief if their child did develop ear pain in the subsequent 12 months.
  Interventions: Other: ear pain counseling
- language power counseling (Active Comparator): The Language Power materials explained the importance of frequent conversations between parents and children and of using encouraging rather than discouraging comments and the PRA reviewed age-appropriate activities in the Learning Games book, and the importance of daily reading using the provided children's book as an example.
  Interventions: Other: language power counseling

INTERVENTIONS:
Other: ear pain counseling — The Ear Pain counseling materials reviewed concepts such as how to recognize ear pain and safely provide pain relief, and how to recognize danger signs that require urgent medical attention. Families were also encouraged to schedule an appointment in the CHC for a possible ear infection rather than going to the emergency department or urgent care facility after hours.
  Arms: ear pain counseling
Other: language power counseling — The Language Power materials explained the importance of frequent conversations between parents and children and of using encouraging rather than discouraging comments and the PRA reviewed age-appropriate activities in the Learning Games book, and the importance of daily reading using the provided children's book as an example.
  Arms: language power counseling

SUMMARY:
Importance: Ear pain is a frequent reason for pediatric visits. Objective: To determine if a program of anticipatory guidance counseling for ear pain at the 12-15 month routine preventive care visit in a predominantly low income population can reduce medical visits to clinic, emergency department (ED), and urgent care (UC).

Design: Single blind randomized control trial of an ear pain counseling program.

Setting: The Child Health Clinic (CHC), a primary care clinic at Children's Hospital Colorado, which serves a predominantly low income population with diverse cultural and ethnic backgrounds.

Participants: 310 mothers were enrolled at their child's 12-15 month well child visit.

Intervention: Structured 10-minute education intervention, given by a research assistant, used a slide presentation that reviewed ear pain Main Outcome and Measures: Number of ED, UC, and clinic visits for otitis media for the 12 month period after entry into the study and whether the visit included a prescription for antibiotics.

DETAILED DESCRIPTION:
The research assistant provided a structured 10 minute education session using 10 PowerPoint slides specific to the subject's assigned group. This was done in the exam room during the child's clinic visit using a portable laptop computer to display the slides, and a copy of the slides was provided to each family at the end of the session.

The Ear Pain counseling materials reviewed concepts such as how to recognize ear pain and safely provide pain relief, and how to recognize danger signs that require urgent medical attention. Families were also encouraged to schedule an appointment in the CHC for a possible ear infection rather than going to the emergency department or urgent care facility after hours. The research assistant provided and reviewed proper dosing instructions for acetaminophen and ibuprofen, and provided a prescription for antipyrine/benzocaine analgesic ear drops to each family to use as pain relief if their child did develop ear pain in the subsequent 12 months.

All participating families completed a demographics survey that included information on race/ethnicity, insurance status, language(s) spoken in the home, and family composition In addition, participants completed the StimQ, the Parent Evaluation of Developmental Status (PEDS), and the he MacArthur-Bates Communicative Development Inventory.

At the child's 24 month preventive care visit, or approximately 12 months after the initial encounter, a research assistant blinded to the participant's study arm assignment met with each family and asked them to once again complete each of the above listed surveys and questionnaires. Those participants who did not present to the CHC for a clinic visit between 24 and 27 months of age, most commonly because they had switched providers or were delayed in scheduling the child's 24 month visit, were contacted by phone and asked to complete the surveys and questionnaires via US mail. If no follow up data had been collected by the time the child reached 30 months of age, that subject was considered lost to follow up.

The electronic medical record (EMR) for each child (EPIC) was reviewed for a diagnosis of otitis media using all otitis related diagnostic codes for 12 months following their initial index visit. The site of each subsequent otitis related visit was documented (CHC, Emergency Department, Urgent care clinic, Ear, Nose and Throat (ENT) clinic) as well as antibiotic that was prescribed. The EMR review documented the number of otitis related visits for each child in total and by site of care as well as the time from the initial index visit to the first otitis related visit with and without an associated antibiotic prescription.

Appropriate statistical tests analyzed differences between study groups and baseline demographic characteristics. Interactions between the study group and dichotomous demographic variables were tested in negative-binomial regression models. When socio-demographic data was missing the enrollee was not included in that sub-analysis. Final stratified regression models represent the relationship between ear pain visits, the study group, and the dichotomous demographic characteristic. Each stratified model was analyzed to represent the appropriate intervention vs. control comparison for each level of the demographic factor [e.g., Post High School education (intervention vs. control) and ≤ High School education (intervention vs. control)].

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12-15 months seen at the CHC for their preventive care visit were eligible for enrollment in the study.

Exclusion Criteria:

* Ventilating tubes
* Down syndrome
* Cardiac disease
* Immunodeficiency disorder
* Family's primary language was something other than English or Spanish

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of Otitis related visits by site of care | 12 months
  The electronic medical record (EMR) for each child (EPIC) was reviewed for a diagnosis of otitis media using all otitis related diagnostic codes for 12 months following their initial index visit.

SECONDARY OUTCOMES:
Time from the initial index visit to the first otitis related visit. | 12 months

OTHER OUTCOMES:
Influence of maternal ethnicity, education, marital status, and age on the effect of ear pain counseling | 12 months
The site of each subsequent otitis related visit was documented (CHC, Emergency Department, Urgent care clinic, ENT clinic). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Berman, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Childrens Hospital Colorado, Aurora, Colorado, United States